CLINICAL TRIAL: NCT06203119
Title: Construction and Clinical Translation of ACE Targeted Nuclear Medicine Imaging Probe
Status: Recruiting | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Hua Zhu, Principal Investigator, Peking University Cancer Hospital & Institute
Other Study IDs: 2023KT160
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Cancer
Keywords: PET/CT; TNBC; 68Ga labeling; diagnosis
MeSH Terms: conditions — Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 68Ga-DOTA-BPP: 68Ga-DOTA-BPP PET/CT: after intravenous injection of 2.96 MBq/ kg body weight of quality-controlled 68Ga-DOTA-BPP, a Siemens Biograph PET/CT scan will be applied within 1 h-2 h, and the scan range will be from the top of the head to 1/3 of the upper thigh.
- 18F-FGD: 18F-FDG PET/CT: after intravenous injection of 2.96 MBq/ kg body weight of quality-controlled 18F-FDG, a Siemens Biograph PET/CT scan will be applied within 1 h, and the scan range will be from the top of the head to 1/3 of the upper thigh.

SUMMARY:
This is an open-label positron emission tomography/computed tomography (PET/CT) study to investigate the clinical predictive value of 68Ga-DOTA-BPP in subjects with triple-negative breast cancer. The visual and semiquantitative methods will be used to assess the PET/CT images

DETAILED DESCRIPTION:
ACE is expressed in triple-negative breast cancer cells. This project develops new type of 68GA-labeled DOTA-BPP, leveraging the inherent strengths of this nuclear medicine discipline, promoted the formulation of the production of this drug To obtain 68Ga-DOTA-BPP injection that can be used in preclinical studies and meets clinical standards. Join a group In clinical patients, 68Ga-DOTA-BPP PET/CT imaging of patients with ACE-positive TNBC was performed, and ACE was obtained To provide evidence for patient screening and efficacy evaluation before targeted therapy with high expression of TNBC, and preliminatively evaluate the level of ACE against high level of ACE. The effect of tumor development can provide a practical basis for the establishment of ACE-targeted PET imaging platform

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old;
2. ECOG score 0 or 1 point;
3. Participants with confirmed TNBC cancer who are suggested by the clinicians to conduct PET/CT imaging for tumor diagnosis or staging.

Exclusion Criteria:

1. Pregnant or nursing;
2. Severe hepatic or renal dysfunction;
3. Low WBC (less than 3 x 10^9/L);
4. Unable to comply with the PET/CT imaging procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Being Cancer Hospital who are confirmed TNBC.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Visual assessment of lesions | 1 year
  Visual analysis of 68Ga-DOTA-BPP PET images will be performed by consensus reading by at least 2 experienced nuclear medicine physician
Semiquantitative assessment of lesions | 1 year
  The standardized uptake values (SUVs) of 68Ga-DOTA-BPP in lesions will be measured by the same nuclear medicine physician for all the cases

SECONDARY OUTCOMES:
ACE expression analysis of tumor tissues | 1 year
  Tumor tissues obtained from biopsy or surgery will be stained for ACE
Correlation analysis of 68Ga-DOTA-BPP uptake and lesion size changes | 1 year
  The SUVs of 68Ga-DOTA-BPP in individual lesions will be compared to the changes in lesion sizes

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics Committee of Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No